CLINICAL TRIAL: NCT02731703
Title: Evaluation of Patient Satisfaction Comparing Conventional, Overdenture and Palateless Overdenture Using Guided Maxillary Implant Placement
Brief Title: Conventional, Overdenture and Palateless Overdenture Oral Health Impact Comparison Study
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-0521
Record Dates: First submitted 2016-03-22; First posted 2016-04-07 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Jaw, Edentulous
Keywords: overdenture; overlay; implant supported; denture; dental prosthesis; maxillary
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Overdenture Treatment: Guided maxillary implant placement with palateless overdenture
  Interventions: Device: Overdenture treatment

INTERVENTIONS:
Device: Overdenture treatment — Conventional, FDA-approved prosthetics will be used in accordance with their labeling and pre-study prescribed standard treatment approach

SUMMARY:
This study will identify and enroll patients already scheduled to receive guided maxillary implant placement with palateless overdenture. Standard clinical practice will be followed for this multi-stage process. The study purpose is to evaluate the degree of satisfaction during the standard progression in order to determine at which post edentulous stage patients achieve maximum satisfaction using the Oral Health Impact Profile 49 (OHIP 49).

DETAILED DESCRIPTION:
The OHIP 49 will be administered at pre-treatment (edentulous condition) and after each visit (i.e., newly fabricated conventional denture, conversion to a 4 implant retained overdenture and finally a 4 implant retained palateless overdenture). Additionally they will be recalled yearly for 5 years.

Participants will have an interim denture fabricated to be worn for 10-12 weeks. During this time, participants will have 4 implants placed and continue wearing the interim denture. At 8 weeks after implant placement, participants will have locator attachments placed on implants and the interim denture snapped into place, termed the 'overdenture.' After 10-12 weeks of wearing this overdenture, patients will receive a new denture, termed 'final palateless overdenture,' which consists of a denture snapped into the 4 implants without a palate. Participants will be evaluated at a 10-12 week followup from insertion of this prosthesis. Participants will complete questionnaires at each stage of treatment.

One year after delivery of the final palateless overdenture and for five consecutive years patients will be asked to return for a follow up appointment.

Estimated duration of patient participation is approximately 5 years and 8 months (271 weeks). Estimated time for active clinical treatment is 8 months (32 weeks) with understanding of flexibility based on laboratory fabricated denture frameworks and adjustments needed for approval of esthetics.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* Able and willing to follow study procedures and instructions
* In good general health
* Edentulous in maxillary arch for a period of at least 6 months
* Have adequate bone volume present to place four maxillary implants without necessity of sinus augmentation or hard and soft tissue grafting ( as determined by the investigator following panoramic radiograph acquisition)

Exclusion Criteria:

* ASA (American Society of Anesthesiologists) Class 3+
* Immunocompromised (Including HIV infection)
* Current drug abuse (self-reported as part of the School of Dentistry health history
* Pregnant or plans to be pregnant at any point during trial
* History of IV or oral bisphosphonate use contraindicating dental implant therapy
* Chronic disease with oral manifestations
* Exhibit Oral pathology
* Ongoing medications initiated less than three months prior to enrollment (medications for chronic medical conditions must be initiated at least three months prior to enrollment.)
* Smoker within the past 6 months
* Diabetes
* Known allergies to any materials used in denture fabrication or implant surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: UNC Graduate Prosthodontics Clinic
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Overall Patient satisfaction OHIP 49 score | End of initial treatment (32 weeks) after all 4 prostheses have each been worn for 10-12 weeks
  The OHIP 49 provides a measure of social impact of oral disorders by providing a comprehensive measure of dysfunction, discomfort and disability resulting from oral cavity conditions. The OHIP 49 is based on the adaptation of the World Health Organization classification. Responses on the OHIP 49 questionnaire are made on a patient satisfaction survey consisting of 49 items organized into 5 subscales (not at all satisfied, not very satisfied, reasonably satisfied, very satisfied, totally satisfied) and responses are based on a Likert scale.

SECONDARY OUTCOMES:
Change in OHIP 49 score of initial edentulous condition to new interim denture | Initial edentulous condition to 10-12 weeks post insertion of new interim denture
  Participant will wear new denture for 10-12 weeks and then OHIP 49 will be administered to compare satisfaction score to their previous edentulous condition.
Change in OHIP 49 score of new interim denture to implant retained interim denture | Interim denture placement to 10-12 weeks post insertion final palateless implant retained overdenture
  Participant will wear implant retained denture for 10-12 weeks and then OHIP 49 will be administered to compare satisfaction score to their previous denture without implant retention.
Change in OHIP 49 score of final palateless implant retained overdenture | 10-12 weeks post insertion of final palateless implant retained overdenture
  Participant will wear final palateless implant retained overdenture for 10-12 weeks and then OHIP 49 will be administered to compare satisfaction score to their previous denture without implant retention.
Change in OHIP 49 score of final palateless implant retained overdenture-Year 1 | 1 Year post insertion of final palateless implant retained overdenture
  Participant will wear final palateless implant retained overdenture for 1 year and then OHIP 49 will be administered to compare satisfaction score to their previous denture without implant retention.
Change in OHIP 49 score of final palateless implant retained overdenture-Year 2 | 2 Year post insertion of final palateless implant retained overdenture
  Participant will wear final palateless implant retained overdenture for 2 years and then OHIP 49 will be administered to compare satisfaction score to their previous denture without implant retention.
Change in OHIP 49 score of final palateless implant retained overdenture-Year 3 | 3 Year post insertion of final palateless implant retained overdenture
  Participant will wear final palateless implant retained overdenture for 3 years and then OHIP 49 will be administered to compare satisfaction score to their previous denture without implant retention.
Change in OHIP 49 score of final palateless implant retained overdenture-Year 4 | 4 Year post insertion of final palateless implant retained overdenture
  Participant will wear final palateless implant retained overdenture for 4 years and then OHIP 49 will be administered to compare satisfaction score to their previous denture without implant retention.
Change in OHIP 49 score of final palateless implant retained overdenture-Year 5 | 5 Year post insertion of final palateless implant retained overdenture
  Participant will wear final palateless implant retained overdenture for 5 years and then OHIP 49 will be administered to compare satisfaction score to their previous denture without implant retention.
Number of participants exhibiting soft tissue complications of final palateless implant retained overdenture | Immediately post insertion of final palateless implant retained overdenture through Year 5
  Participant will return yearly for 5 years to evaluate possible complications in regards to health of soft tissue
Number of participants exhibiting fit complications of final palateless implant retained overdenture | Immediately post insertion of final palateless implant retained overdenture through Year 5
  Participant will return yearly for 5 years to evaluate possible complications in regards to the fit of the palateless implant retained overdenture
Number of participants exhibiting retention complications of final palateless implant retained overdenture | Immediately post insertion of final palateless implant retained overdenture through Year 5
  Participant will return yearly for 5 years to evaluate possible complications in regards to the retention of the palateless implant retained overdenture

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg De Kok, DDS MS, Principal Investigator — Associate Professor UNC School of Dentistry
Locations (1):
- University of North Carolina School of Dentistry, Graduate Prosthodontics, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albrektsson T, Zarb G, Worthington P, Eriksson AR. The long-term efficacy of currently used dental implants: a review and proposed criteria of success. Int J Oral Maxillofac Implants. 1986 Summer;1(1):11-25. No abstract available. PMID 3527955
- [Background] Arisan V, Karabuda CZ, Ozdemir T. Implant surgery using bone- and mucosa-supported stereolithographic guides in totally edentulous jaws: surgical and post-operative outcomes of computer-aided vs. standard techniques. Clin Oral Implants Res. 2010 Sep;21(9):980-8. doi: 10.1111/j.1600-0501.2010.01957.x. Epub 2010 May 24. PMID 20497439
- [Background] Bragger U. Radiographic parameters: biological significance and clinical use. Periodontol 2000. 2005;39:73-90. doi: 10.1111/j.1600-0757.2005.00128.x. No abstract available. PMID 16135065
- [Background] Branemark PI, Hansson BO, Adell R, Breine U, Lindstrom J, Hallen O, Ohman A. Osseointegrated implants in the treatment of the edentulous jaw. Experience from a 10-year period. Scand J Plast Reconstr Surg Suppl. 1977;16:1-132. No abstract available. PMID 356184
- [Background] Cardelli P, Cecchetti F, Montani M, Bramanti E, Arcuri C. Clinical assessment of submerged vs non-submerged implants placed in pristine bone. Oral Implantol (Rome). 2014 May 19;6(4):89-93. eCollection 2013 Apr. PMID 24971162
- [Background] Cavallaro JS Jr, Tarnow DP. Unsplinted implants retaining maxillary overdentures with partial palatal coverage: report of 5 consecutive cases. Int J Oral Maxillofac Implants. 2007 Sep-Oct;22(5):808-14. PMID 17974117
- [Background] Cranin AN, DeGrado J, Kaufman M, Baraoidan M, DiGregorio R, Batgitis G, Lee Z. Evaluation of the Periotest as a diagnostic tool for dental implants. J Oral Implantol. 1998;24(3):139-46. doi: 10.1563/1548-1336(1998)0242.3.CO;2. PMID 9893520
- [Background] Feine JS, Carlsson GE, Awad MA, Chehade A, Duncan WJ, Gizani S, Head T, Lund JP, MacEntee M, Mericske-Stern R, Mojon P, Morais J, Naert I, Payne AG, Penrod J, Stoker GT, Tawse-Smith A, Taylor TD, Thomason JM, Thomson WM, Wismeijer D. The McGill consensus statement on overdentures. Mandibular two-implant overdentures as first choice standard of care for edentulous patients. Montreal, Quebec, May 24-25, 2002. Int J Oral Maxillofac Implants. 2002 Jul-Aug;17(4):601-2. No abstract available. PMID 12182304
- [Background] Fortin T, Bosson JL, Isidori M, Blanchet E. Effect of flapless surgery on pain experienced in implant placement using an image-guided system. Int J Oral Maxillofac Implants. 2006 Mar-Apr;21(2):298-304. PMID 16634502
- [Background] Fransson C, Lekholm U, Jemt T, Berglundh T. Prevalence of subjects with progressive bone loss at implants. Clin Oral Implants Res. 2005 Aug;16(4):440-6. doi: 10.1111/j.1600-0501.2005.01137.x. PMID 16117768
- [Background] Gendreau L, Loewy ZG. Epidemiology and etiology of denture stomatitis. J Prosthodont. 2011 Jun;20(4):251-60. doi: 10.1111/j.1532-849X.2011.00698.x. Epub 2011 Apr 4. PMID 21463383
- [Background] Heitz-Mayfield LJ. Peri-implant diseases: diagnosis and risk indicators. J Clin Periodontol. 2008 Sep;35(8 Suppl):292-304. doi: 10.1111/j.1600-051X.2008.01275.x. PMID 18724857
- [Background] Nilsson B. The occurrence of taste buds in the palate of human adults as evidenced by light microscopy. Acta Odontol Scand. 1979;37(5):253-8. doi: 10.3109/00016357909004694. PMID 294117
- [Background] Pjetursson BE, Asgeirsson AG, Zwahlen M, Sailer I. Improvements in implant dentistry over the last decade: comparison of survival and complication rates in older and newer publications. Int J Oral Maxillofac Implants. 2014;29 Suppl:308-24. doi: 10.11607/jomi.2014suppl.g5.2. PMID 24660206
- [Background] Roos-Jansaker AM, Lindahl C, Renvert H, Renvert S. Nine- to fourteen-year follow-up of implant treatment. Part II: presence of peri-implant lesions. J Clin Periodontol. 2006 Apr;33(4):290-5. doi: 10.1111/j.1600-051X.2006.00906.x. PMID 16553638
- [Background] Santos BF, dos Santos MB, Santos JF, Marchini L. Patients' Evaluations of Complete Denture Therapy and Their Association with Related Variables: A Pilot Study. J Prosthodont. 2015 Jul;24(5):351-7. doi: 10.1111/jopr.12286. Epub 2015 Apr 9. PMID 25864962
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981
- [Background] Vercruyssen M, Cox C, Coucke W, Naert I, Jacobs R, Quirynen M. A randomized clinical trial comparing guided implant surgery (bone- or mucosa-supported) with mental navigation or the use of a pilot-drill template. J Clin Periodontol. 2014 Jul;41(7):717-23. doi: 10.1111/jcpe.12231. Epub 2014 Apr 10. PMID 24460748
- [Background] Wang F, Monje A, Huang W, Zhang Z, Wang G, Wu Y. Maxillary Four Implant-retained Overdentures via Locator(R) Attachment: Intermediate-term Results from a Retrospective Study. Clin Implant Dent Relat Res. 2016 Jun;18(3):571-9. doi: 10.1111/cid.12335. Epub 2015 Mar 23. PMID 25810348
- [Background] Zembic A, Tahmaseb A, Wismeijer D. Within-Subject Comparison of Maxillary Implant-Supported Overdentures with and without Palatal Coverage. Clin Implant Dent Relat Res. 2015 Jun;17(3):570-9. doi: 10.1111/cid.12125. Epub 2013 Jul 30. PMID 23899103
- [Background] Zitzmann NU, Berglundh T. Definition and prevalence of peri-implant diseases. J Clin Periodontol. 2008 Sep;35(8 Suppl):286-91. doi: 10.1111/j.1600-051X.2008.01274.x. PMID 18724856
- [Background] Zitzmann NU, Marinello CP. Treatment outcomes of fixed or removable implant-supported prostheses in the edentulous maxilla. Part II: clinical findings. J Prosthet Dent. 2000 Apr;83(4):434-42. doi: 10.1016/s0022-3913(00)70038-2. PMID 10756293
- [Background] Roos J, Sennerby L, Lekholm U, Jemt T, Grondahl K, Albrektsson T. A qualitative and quantitative method for evaluating implant success: a 5-year retrospective analysis of the Branemark implant. Int J Oral Maxillofac Implants. 1997 Jul-Aug;12(4):504-14. PMID 9274079